CLINICAL TRIAL: NCT02972606
Title: Online Psychological Treatment for People With Painful HIV-related Peripheral Neuropathy (OPEN Study): Qualitative Investigation of Treatment Needs
Brief Title: OPEN Study: Pain Management Treatment Needs Interviews
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Imperial College London (Other); Chelsea and Westminster NHS Foundation Trust (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 205949
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2016-09

CONDITIONS: HIV; Peripheral Neuropathy
Keywords: HIV; Peripheral Neuropathy; Chronic Pain; Qualitative Research
MeSH Terms: conditions — Peripheral Nervous System Diseases; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Presently, there are few options for medically managing HIV-related painful peripheral sensory neuropathy (HIV-SN). Psychological treatments, including Cognitive Behavioural Therapy (CBT), represent a potentially viable addition to the treatment of painful HIV-SN. However, there is a scarcity of research on psychological treatment approaches for pain management in people with HIV. This study will use in-depth semi-structured interviews to examine the needs of people with painful HIV-SN for a psychologically-based pain management treatment that may be delivered over the Internet. Interview questions will examine participants' needs in terms of treatment content and delivery format. Men and women, ethnic minorities, and people who use recreational drugs will be sampled to ensure that interview responses reflect the views of people most commonly suffering from this condition. Approximately 30 people will be recruited for the study. The interviews will be audio recorded, transcribed verbatim, and coded to identify themes. The interview responses will be used to develop and tailor a version of CBT for people with painful HIV-SN. It is hoped that tailoring the treatment based on the qualitative interview responses will increase the acceptability of the treatment and will improve treatment adherence rates for a future study.

DETAILED DESCRIPTION:
This report is independent research supported by the National Institute for Health Research (NIHR Post Doctoral Fellowship, Dr Whitney Scott, PDF-2015-08-059). The views expressed in this publication are those of the authors and not necessarily those of the NHS, the National Institute for Health Research or the Department of Health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Living with HIV.
* A positive screen for peripheral sensory neuropathy, as indicated by: presence of self-reported bilateral foot pain and/or numbness in a symmetrical distribution.
* Positive screen for symptoms of neuropathic pain in the feet, as indicated by a score of greater than or equal to 3 on the patient reported outcomes section of the Neuropathic Pain Interview.
* Pain in the feet present most days for at least 3 months.
* Average pain intensity of greater than or equal to 4/10.
* Average interference of pain with daily activities is greater than or equal to 4/10.

Exclusion Criteria:

* Presence of excessive alcohol consumption, hypothyroidism, vitamin B12 deficiency, diabetes, exposure to isoniazid or chemotherapy drug treatment, or a known history of a neuropathy due to a cause other than HIV or antiretroviral treatment
* Unable to conduct interview in English.
* Current diagnosis of dementia or learning disability.
* Unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with HIV and painful peripheral neuropathy. We will purposively sample men, women, ethnic minorities, and people who use recreational drugs .
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Scott, PhD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - King's College London, London
  - Chelsea & Westminster Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott W, Garcia Calderon Mendoza Del Solar M, Kemp H, McCracken LM, C de C Williams A, Rice ASC. A qualitative study of the experience and impact of neuropathic pain in people living with HIV. Pain. 2020 May;161(5):970-978. doi: 10.1097/j.pain.0000000000001783. PMID 31855944
- See also: Published peer-reviewed paper — https://journals.lww.com/pain/Abstract/publishahead/A_qualitative_study_of_the_experience_and_impact.98522.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With HIV and Neuropathy: Participants with HIV and Neuropathy (this was a qualitative study and participants were not assigned to arms).
Period: Overall Study
Arm/Group | Participants With HIV and Neuropathy
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis.
Groups:
- Participants With HIV and Neuropathy: Participants with HIV and Neuropathy who completed semi-structured interviews.
Arm/Group | Participants With HIV and Neuropathy
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White British/European | 17
  Race/Ethnicity: Black British/African | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed a Semi-Structure Interview
Description: Semi-structured interview performed at one occasion where the patient describes his/her experience living with painful peripheral neuropathy and his/her thoughts about a psychological treatment for managing pain.
Time Frame: Day 1
Population: All participants were analysed
Measure: Count of Participants; unit: Participants
Groups:
- Not Applicable: Not applicable as this is a qualitative study
Arm/Group | Not Applicable
Number analyzed (Participants) | 26
Participants | 26

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not recorded. There was a risk management procedure that involved contacting the participants' GP if clinically meaningful distress or other symptoms were identified during the qualitative interviews. However, the frequency of contacting GPs to manage this risk was not systematically recorded as this was not an intervention study.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not recorded. There was a risk management procedure that involved contacting the participants' GP if clinically meaningful distress or other symptoms were identified during the qualitative interviews. However, the frequency of contacting GPs to manage this risk was not systematically recorded as this was not an intervention study.
Groups:
- EG000: Not applicable. This is a qualitative study.
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02972606/Prot_SAP_000.pdf